CLINICAL TRIAL: NCT03389269
Title: Investigation of Acute Physiological Effects of Aspiration Therapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Christina Charlotte Nexoe-Larsen, MD, pH.D student, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-16038453
Record Dates: First submitted 2017-11-28; First posted 2018-01-03 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — Gastric content postprandial. Plasma and serum. Urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Obese patients treated with AspireAssist: Healthy, obese with BMI > 27, treated with AspireAssist for weight management, the postprandial glucose metabolism will be tested with a meal test
  Interventions: Other: Meal test
- Matched controls: Healthy, obese with BMI > 27, the postprandial glucose metabolism will be tested with a meal test
  Interventions: Other: Meal test

INTERVENTIONS:
Other: Meal test — 240 min mixed meal test with aspiration using AspireAssist.

SUMMARY:
In the present study, the investigators aim to investigate postprandial physiology in patients who have had the Aspire Assist® inserted. This will involve a standardised mixed meal test (MMT) with subsequent aspiration of gastric content compared to MMT without aspiration. Furthermore, a comparison will be made between the aspiration group and a control group in order to evaluate whether continuous treatment with aspiration therapy affect the postprandial physiology. The primary outcomes of the trial are differences in postprandial plasma/serum glucose, insulin and gut hormone excursions during MMT with and without aspiration. Secondary outcomes encompass evaluation of satiety, gastric emptying and gallbladder motility following MMT with and without aspiration. Also, food intake during a subsequent ad libitum meal will be evaluated.

DETAILED DESCRIPTION:
It is generally agreed that the increasing incidence of obesity mainly is caused by the adoption of a sedentary lifestyle combined with excessive caloric intake. So far, preventive measures and interventions based on lifestyle modifications have not been able to affect the western lifestyle to a degree that remedies the increasing prevalence of obesity. Likewise, no medical interventions have yet been able to induce and maintain significant major weight loss in obese populations. In contrast, bariatric surgery prompts a significant and often sustained weight loss, which frequently triggers remission of obesity-related comorbidities. However, bariatric surgery is invasive, irreversible and costly. Aspiration therapy was introduced as a less invasive and cheaper treatment for obesity. According to some studies, aspiration therapy is nearly as effective as Roux-en-Y gastric bypass in terms of excess weight loss after one year. Thus, aspiration therapy may aspire as an alternative treatment option for obesity with lower risk of complications than bariatric surgery.

The risk of developing impaired glucose tolerance and overt type 2 diabetes rises along with increasing obesity. The estimated risk of developing type 2 diabetes increases 3-fold with a body mass index (BMI) of 25-29.9 kg/m2 (overweight) and ~20-fold with a BMI >35 kg/m2 (severely obese) compared to a normal BMI (<25 kg/m2) (6). Type 2 diabetes is a complex, multi-organ metabolic disorder and is associated with serious complications, reduced quality of life and early death. The disease is characterized by hyperglycaemia and, thus, elevated haemoglobinA1c (HbA1c) (>6.5% or >48mmol/mol), which is a blood parameter used clinically as a measure of mean blood glucose over time (~3 months). Studies have shown that up to 70% of the mean plasma glucose levels is caused by postprandial plasma glucose excursions. Moreover, postprandial hyperglycaemia in itself seems to be associated with an elevated risk of cardiovascular disease due to unfavourable effect on both small and large blood vessels. Accordingly, postprandial hyperglycaemia has been suggested to constitute a better predictor of mortality risk than fasting plasma glucose concentrations in both patients with type 2 diabetes and individuals with normal glucose tolerance. Since the prevalence of impaired glucose tolerance is ~2-fold higher in obese compared to lean individuals, postprandial hyperglycaemia poses a great risk of developing severe comorbidities such as cardiovascular disease and type 2 diabetes for obese individuals and may increase mortality in this group. It is yet unknown whether aspiration therapy can attenuate the plasma glucose response to a meal. Due to the reduced amount of food reaching the intestine after aspiration, it seems likely that aspiration therapy reduces postprandial plasma glucose excursions and thereby prevents potential postprandial hyperglycaemia.

It is well known that an orally administered glucose load elicits a greater insulin secretion response compared to an intravenous infusion of glucose resulting in identical plasma glucose elevations. This phenomenon is called the incretin effect. The incretin effect is primarily driven by the insulinotropic gut hormones glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP). These so-called incretin hormones play crucial roles in regulation of glucose homeostasis and appetite. GLP-1 is produced in the intestinal mucosa by the so-called enteroendocrine L cells, which are predominantly localised in the distal part of the small intestine and the colon. GIP originates from enteroendocrine K 5 cells in the gut mucosa. K cells are assumed to be predominant in the proximal part of the small intestine. Both GLP-1 and GIP are secreted in response to ingestion of nutrients and have strong glucose-dependent insulinotropic effects on pancreatic beta cells. The incretin hormones are of interest in the present study, because impaired incretin effect is an early sign of dysmetabolism in obese individuals and a distinctive feature of type 2 diabetes, suggesting that the impaired glucose tolerance of these patients is, at least in part, due to a defective incretin system. Whether aspiration of gastric content after a meal affects postprandial incretin hormone response has not been elucidated. The investigators plan to investigate meal-induced incretin hormone excursions in plasma with and without aspiration therapy and compare the results to a matched control group.

In addition to GLP-1 and GIP, several other gut-related hormones are known to regulate glucose homeostasis and appetite. Glucagon is a peptide hormone secreted from the pancreatic alpha cells. Glucagon acts opposite to insulin by promoting hepatic gluconeogenesis and glycogenolysis causing increased plasma glucose concentrations. Oxyntomodulin and pancreatic peptide YY3-36 (PYY) are peptide hormones secreted by the enteroendocrine L cells in response to feeding and both suppress appetite. Gastrin is a hormone secreted by G cells localised in the pyloric antrum, duodenum and pancreas. Gastrin stimulates acid (HCl) secretion and gastric emptying by increasing gastric motility. Cholecystokinin (CCK) is a peptide hormone secreted by the enteroendocrine I cells in the duodenum. CCK promotes bile release from the gallbladder and also acts as an appetite suppressant. To this point, it is unknown how aspiration therapy affects these appetite- and glucose-regulating hormones during a meal. The investigators aim to investigate this during standardised mixed meal tests with and without aspiration.

Furthermore, it is relevant to examine the effect of aspiration therapy on satiety. Thus, the investigators aim to evaluate the effect of aspiration therapy on satiety before, during and after a mixed meal as well as food intake after the MMT with and without aspiration evaluated through an ad libitum meal provided at the end of the experimental days.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have had the Aspire Assist inserted (the aspiration therapy group)
* Age between 18-75 years
* Able to understand written patient information and sign informed consent

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Severe comorbidities that, at the discretion of the investigators, exclude study participation (e.g. chronic obstructive pulmonary disease (COPD) stage III, significant cardiac arrhythmias etc.)
* Previous gastrointestinal surgery (excluding cholecystectomy and appendectomy)
* Gastrointestinal conditions making the participant unsuitable for participation (e.g. ulcerative colitis, Crohn´s disease, clinically significant food allergies, candidiasis etc.)
* Anaemia with a haemoglobin value <6.2 mmol/l (<10 g/dl) for women and <7.4 mmol/l (< 12 g/dl) for men at time of screening
* Abuse of alcohol and/or drugs, or any other co-existing conditions that will make the participant unsuitable to attend to the study schedule, as deemed by the investigators
* Pregnancy or desire to become pregnant during the study period
* Exceptional conditions which, at the discretion of the investigators, preclude the participation in the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: It is planned to recruit up to 25 patients who have had the Aspire Assist inserted. Furthermore, 10 healthy control participants matched for age, weight, height, BMI and sex will be recruited
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Plasma glucose concentration | 0-240 min
  mmol/l, collected during mixed meal test and analysed by YSI STAT 2300

SECONDARY OUTCOMES:
Serum Insulin | 0-240 min
  pmol/l, Collected during mixed meal test
plasma GLP-1 | 0-240 min
  pmol/l, Collected during mixed meal test
Indirect Calorimetry | 0-240 min
  Resting metabolic rate measured by O2 consumption during mixed meal test
Gallbladder volume | 0-240 min
  Measured during mixed meal test by UL and calculated by this equation: π/6*D1*D2*D3/1000, D1 = longitudinal diameter, D2 = cross section width, D3 = cross sectional width
Ad libitum meal intake | 30 min
  post meal test
Appetite | 0-240 min
  Evaluated by visual analogue scale (VAS 0-10, where 0 is no appetite and 10 is very hungry) during mixed meal test
Plasma GLP-2 | 0-240 min
  pmol/l, Collected during mixed meal test
Plasma GIP | 0-240 min
  pmol/l, Collected during mixed meal test
Plasma Glucagon | 0-240 min
  pmol/l, Collected during mixed meal test
Plasma PYY | 0-240 min
  pmol/l, Collected during mixed meal test
Plasma Oxyntomodulin | 0-240 min
  pmol/l, Collected during mixed meal test
plasma ghrelin | 0-240 min
  pmol/l, Collected during mixed meal test
Plasma acetaminophen | 0-240 min
  mmol/L, Collected during mixed meal test
plasma c-peptide | 0-240 min
  pmol/l, Collected during mixed meal test
Plasma CCK | 0-240 min
  pmol/l, Collected during mixed meal test
plasma gastrin | 0-240 min
  pmol/l, Collected during mixed meal test

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, Proff, Principal Investigator — Center for diabetes research, gentofte hospital
Locations (1):
- Center for Diabetes Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No